CLINICAL TRIAL: NCT04360512
Title: Dose-response of Posterior Talus Mobilizations on Ankle Range of Motion and Overall Mobility in Older Adults
Brief Title: Dose-response of Talus Mobilizations
Acronym: ANKLE_ROM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended due to the covid-19 pandemic.
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández, PT, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DHG05
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Aging Problems
Keywords: ROM; Manual therapy; Dose-response; Mobilization; Ankle

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- One session (Experimental): One session of talus posteriorization
  Interventions: Procedure: Posteriorization of the talus
- Two sessions (Experimental): Two sessions of talus posteriorization
  Interventions: Procedure: Posteriorization of the talus
- Three sessions (Experimental): Three sessions of talus posteriorization
  Interventions: Procedure: Posteriorization of the talus
- Four sessions (Experimental): Four sessions of talus posteriorization
  Interventions: Procedure: Posteriorization of the talus

INTERVENTIONS:
Procedure: Posteriorization of the talus — Three sets of a 30-s grade IV mobilization

SUMMARY:
Ankle mobility limitations are common in older adults. A possible treatment to restore joint mobility is manual therapy based on mobilization techniques, in this case, applied on the ankle joint. Previous research had proposed different treatment volumes (one to twelve sessions), but shown a different and non-consistent degree of effectiveness according to such factor. Therefore, this work aims to determine the dose-response relationship of manual therapy (talus mobilizations) on ankle range of motion in the older adult. Secondarily, this research will appraise whether a likely improvement in ankle mobility may have an impact on the overall mobility (i.e. gait, get up from a chair).

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults
* Over 60 years
* Limited ankle dorsiflexion range of motion

Exclusion Criteria:

* Not willing to participate or signing a consent form
* Lower limb injury in the three months prior to the study (ex. sprain)
* Diagnosed condition that may influence mobility assessments (i.e. stroke)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Treatment dose | Change from baseline to end of intervention (2 weeks)
  Number of sessions of experimental intervention needed to induce a clinically important gain in ankle mobility after the intervention. A baseline progression over 4.6º in the Lunge test will be considered clinically important (Powden, 2015), so that the number of sessions will be established when this threshold is exceeded (see secondary outcome) .

SECONDARY OUTCOMES:
The Lunge test | Change from baseline, to end of intervention (2 weeks) and follow-up (10 weeks)
  Weight bearing ankle dorsiflexion range of motion. This test will measure the maximum tilt of the tibia that a subject can perform while standing and bearing the weight on the limb without lifting the heel from the floor. A Baseline® Digital Inclinometer (Fabrication Enterprises Inc) will be used to assessed this outcome. Values below 35º indicate limited mobility. A baseline progression over 4.6º will be considered clinically important (Powden, 2015). This mobility gain will be used to determine the dose-response relationship: number of sessions of talus mobilizations needed to induce a clinically important gain in ankle mobility after the intervention (see primary outcome measure)
Active ankle range of motion | Change from baseline, to end of intervention (2 weeks) and follow-up (10 weeks)
  Non-weight bearing active ankle range of motion in the sagittal plane: dorsi to plantarflexion full range of motion. This will be assessed with a telescopic goniometer, with the participant laying in supine with a wedge under the knees to eliminate the tension of the gastrocnemius muscles. Values below 59º indicate limited ankle mobility. The minimal detectable change for this measure has not been well established in literature. A baseline progression over 5.2º will be considered clinically important (Searle, 2018; Konor, 2012)
Timed up and go test (TUG) | Change from baseline, to end of intervention (2 weeks) and follow-up (10 weeks)
  A timed test used to assess overall mobility and dynamic balance, in which the time taken to get up from and arm-chair, walk three meters, turn around a cone and come back to sit again, is registered to estimate the functional mobility. We will consider times below 12 s as normal performances in the study populattion, and below 13,5 s as low risk of falling. A baseline change over 2.08 s will be considered clinically important (Donoghue, 2019)

OTHER OUTCOMES:
Euro Quality of Life Five Dimensions (EQ-5D) | Change from baseline, to follow-up (10 weeks)
  The descriptive system comprises five dimensions to assess health related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state

CONTACTS AND LOCATIONS:
Overall Officials: José-María Blasco, PT, PhD, Study Director — University of Valencia; David Hernández-Guillén, PT, PhD, Study Chair — University of Valencia; Catalina Tolsada-Velasco, PT, Principal Investigator — University of Valencia
Locations (1):
- Universidad de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided